CLINICAL TRIAL: NCT05911724
Title: Diagnostic and Prognostic Roles of Inflammatory Biomarkers in Coronary Heart Disease and Heart Failure Patients Treated With Empagliflozin.
Brief Title: Association Between Inflammatory Biomarkers in CVD Patients on Empagliflozin.
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Other Study IDs: inflammatory biomarkers in CVD
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Stable Angina; Heart Failure
Keywords: vaspin; visfatin; lipoprotein A; high-sensitivity C-reactive protein; sortilin; homocysteine; troponin I; fetuin A
MeSH Terms: conditions — Angina, Stable; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 60 Healthy Subjects.
  Interventions: Other: Group I Healthy
- Group II: 60 Patients with Stable Angina on empagliflozin 10 mg once daily for 6 months before the beginning of the study.
  Interventions: Drug: CAD-Empagliflozin 10 mg once daily for 6 months before the beginning of the study
- Group III: 60 Patients with Heart Failure on empagliflozin 10 mg once daily for 6 months before the beginning of the study.
  Interventions: Drug: HF-Empagliflozin 10 mg once daily for 6 months before the beginning of the study

INTERVENTIONS:
Other: Group I Healthy — Healthy Subjects
  Groups: Group I
Drug: CAD-Empagliflozin 10 mg once daily for 6 months before the beginning of the study — Group II: Stable Angina Patients
  Other Names: Empa- CAD
  Groups: Group II
Drug: HF-Empagliflozin 10 mg once daily for 6 months before the beginning of the study — Group III: Heart Failure Patients
  Other Names: Empa-HF
  Groups: Group III

SUMMARY:
The association of novel inflammatory biomarkers with cardiovascular diseases is still obscure. The present study aimed to investigate the relationship of various inflammatory biomarkers with the existence as well as the extent of heart failure (HF) and coronary artery disease (CAD), suggesting a link between inflammation and cardiovascular diseases and all-cause 30- and -90 day of hospital readmission. Methods: We enrolled a total of 120 patients with HF, asymptomatic CAD and 60 healthy controls (HC) without cardiovascular diseases.

DETAILED DESCRIPTION:
* The present study aimed to investigate the relationship of various inflammatory biomarkers with the existence as well as the extent of heart failure (HF) and coronary artery disease (CAD), suggesting a link between inflammation and cardiovascular diseases and all-cause 30- and -90 day of hospital readmission in patients on empagliflozin 10 mg once daily for 6 months before the beginning of the study.
* We enrolled a total of 60 patients with HF, 60 asymptomatic CAD patients and 60 healthy controls (HC) without cardiovascular diseases.

Group I: 60 Healthy Subjects. Group II: 60 Patients with Stable Angina (asymptomatic CAD). Group III: 60 Patients with Heart Failure.

* Clinical parameters, glycemic and lipid profile, vaspin, visfatin, high-sensitivity C-reactive protein, sortilin, homocysteine, troponin I, fetuin A and lipoprotein A levels were assayed.
* Patients will be followed up to assess all-cause 30- and -90 day of hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* Either sex, aged 18 years or older.
* new-onset AHF or acute decompensation of chronic HF,
* CAD (including previous myocardial infarction, previous percutaneous or surgical coronary revascularization, or angiographic evidence that one or more major coronary arteries had narrowed by 50% or more).
* On empagliflozin 10 mg once daily for 6 months before the beginning of the study.

Exclusion Criteria:

* severe liver/
* kidney dysfunction;
* severe systemic disease (such as the diseases of respiratory system/ digestive system/ nervous system etc.);
* malignant tumor;
* acute/ chronic infectious diseases;
* autoimmune disease or connective tissue disease;
* major trauma or surgical operation over the past three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group I: 60 Healthy Subjects. Group II: 60 Patients with Stable Angina (asyptomatic CAD), on empagliflozin 10 mg once daily for 6 months before the beginning of the study.
  Group III: 60 Patients with Heart Failure, on empagliflozin 10 mg once daily for 6 months before the beginning of the study.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
All Cause 30 day hosptial admission | 1 month
  Number of patients admited to hospital during 1 month.
All Cause 90 day hosptial admission | 3 months
  Number of patients admited to hospital during 3 month.
vaspin (ng/ml) | 1 month
  vaspin blood concentration
visfatin (ng/ml) | 1 month
  visfatin blood concentration
Sortillin (pg/ml) | 1 month
  Sortillin blood concentration
Homocystien(umol/L) | 1 Month
  Homocystien blood concentration
Troponin.I (ng/ml) | 1 Month
  Troponin.I blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ibtsam Khairat, Ass. Prof., Study Director — Tanta University; Ahmed A. El-Sherbeni, Lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konig P, Mayer O, Bruthans J, Seidlerova J, Materankova M, Gelzinsky J, Rychecka M, Karnosova P, Wohlfahrt P, Cifkova R, Filipovsky J. The prognostic importance of subclinical heart failure in stable coronary heart disease patients. Acta Cardiol. 2020 Aug;75(4):329-336. doi: 10.1080/00015385.2019.1590958. Epub 2019 Apr 3. PMID 30942129
- [Background] Eisen A, Benderly M, Behar S, Goldbourt U, Haim M. Inflammation and future risk of symptomatic heart failure in patients with stable coronary artery disease. Am Heart J. 2014 May;167(5):707-14. doi: 10.1016/j.ahj.2014.01.008. Epub 2014 Feb 22. PMID 24766981
- [Background] Held C, White HD, Stewart RAH, Budaj A, Cannon CP, Hochman JS, Koenig W, Siegbahn A, Steg PG, Soffer J, Weaver WD, Ostlund O, Wallentin L; STABILITY Investigators. Inflammatory Biomarkers Interleukin-6 and C-Reactive Protein and Outcomes in Stable Coronary Heart Disease: Experiences From the STABILITY (Stabilization of Atherosclerotic Plaque by Initiation of Darapladib Therapy) Trial. J Am Heart Assoc. 2017 Oct 24;6(10):e005077. doi: 10.1161/JAHA.116.005077. PMID 29066452
- [Background] Papaioannou V, Pneumatikos I, Maglaveras N. Association of heart rate variability and inflammatory response in patients with cardiovascular diseases: current strengths and limitations. Front Physiol. 2013 Jul 10;4:174. doi: 10.3389/fphys.2013.00174. eCollection 2013. PMID 23847549
- [Background] Williams ES, Shah SJ, Ali S, Na BY, Schiller NB, Whooley MA. C-reactive protein, diastolic dysfunction, and risk of heart failure in patients with coronary disease: Heart and Soul Study. Eur J Heart Fail. 2008 Jan;10(1):63-9. doi: 10.1016/j.ejheart.2007.11.003. Epub 2007 Dec 21. PMID 18160340
- [Derived] El-Sherbeni AA, Khedr NF, Khairat I, Werida RH. Diagnostic and Prognostic Roles of Inflammatory Biomarkers in Patients With Coronary Heart Disease and Heart Failure Treated With Empagliflozin. Clin Ther. 2025 Aug;47(8):e1-e11. doi: 10.1016/j.clinthera.2025.04.019. Epub 2025 May 24. PMID 40413121